CLINICAL TRIAL: NCT04203186
Title: A Phase 1 Clinical Trial To Evaluate The Safety and Infectivity Of Direct Venus Inoculation of Aseptic, Purified, Cryopreserved Plasmodium Falciparum 7G8 And NF54 Challenge Strains (PfSPZ) in a Head-To-Head Comparative Study
Brief Title: A Clinical Trial to Evaluate Plasmodium Falciparum 7G8 and NF54 Challenge Strains (PfSPZ) in a Head-to-head Comparative Study - (ECG-CHMI)
Acronym: ECG-CHMI
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Funding was lost due to the COVID19 Pandemic
Sponsor: U.S. Army Medical Research and Development Command (U.S. Federal Agency)
Collaborators: Naval Medical Research Center (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Diagnostic
Other Study IDs: 19239
Record Dates: First submitted 2019-12-16; First posted 2019-12-18 (Actual); Last update posted 2020-05-08 (Actual); Status verified 2020-05

CONDITIONS: Plasmodium Falciparum
MeSH Terms: conditions — Malaria, Falciparum | interventions — atovaquone, proguanil drug combination; Artemether; Lumefantrine; Artemether, Lumefantrine Drug Combination

STUDY DESIGN:
Intervention Model Description: 2 parallel test groups to directly compare clinical and laboratory characteristics
Who Masked: Participant, Care Provider, Investigator
Masking Description: double-blind, randomized, placebo-controlled trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 - PfSPZ, (NF54) strain (Active Comparator): Group 1 (N=9) will receive PfSPZ Challenge (NF54) A one-time dose of 3,200 aseptic, purified, cryopreserved, non-attenuated Plasmodium falciparum (Pf) NF54 sporozoites (Pf SPZ Challenge) Mode of administration: Direct venous inoculation (DVI) through a 25 gauge needle and syringe
  Interventions: Drug: atovaquone-proguanil
- Group 2 - PfSPZ, (7G8) strain (Active Comparator): Group 2 (N=9) will receive PfSPZ Challenge (7G8) A one-time dose of 3,200 aseptic, purified, cryopreserved, non-attenuated Plasmodium falciparum 7G8 sporozoites (Pf SPZ Challenge) Mode of administration: Direct venous inoculation (DVI) through a 25 gauge needle and syringe
  Interventions: Drug: atovaquone-proguanil

INTERVENTIONS:
Drug: atovaquone-proguanil — Malaria standard treatment regimen
  Other Names: artemether/lumefantrine (AL; Coartem)

SUMMARY:
A comparison of Malaria events (symptoms and signs of malaria) experienced by subjects infected with PfSPZ Challenge (NF54) vs. PfSPZ Challenge (7G8).

DETAILED DESCRIPTION:
The single center study is designed as a double-blind, randomized, placebo-controlled CHMI trial with 2 parallel test groups to directly compare clinical and laboratory characteristics of the NF54 and 7G8 strains of PfSPZ Challenge. This study will also evaluate signatures of and time to parasitemia by multiple methods and evaluate physiologic status data collected by non-invasive wearable monitors before and during Plasmodium falciparum infection to characterize and trend physiologic changes appearing prior to the onset of parasitemia.

PfSPZ Challenge (aseptic, purified, cryopreserved, infectious Plasmodium falciparum sporozoites) or normal saline will be administered by direct venous inoculation (DVI) by 25-gauge needle and syringe to healthy malaria naïve adults.

Data generated from samples collected for biomarker assay analysis will be useful for developing predictive models to evaluate the efficacy of malaria vaccine candidates.

ELIGIBILITY:
Inclusion Criteria:

* Adults (male or non-lactating, non-pregnant female)
* Between the ages of 18 and 45 (inclusive) at the time of enrollment
* Body weight equal to or greater than 110 lbs
* Available and willing to participate for duration of study
* Able and willing to provide a written informed consent
* Able to complete an Assessment of Understanding with a score of at least 80% correct
* In good general health with no clinically significant health problems as established by medical history, physical examination, and laboratory screening
* Sexually active females, unless surgically sterile or at least 1 year post-menopausal, must use an effective method of avoiding pregnancy (Section 5.4.5.3) from 14 days prior to CHMI and agree to continue using such precautions during the study until at least 2 months after CHMI
* If female subjects are unable to bear children due to menopause or have had a procedure performed (e.g. tubal ligation or hysterectomy), a medical note from a physician is required
* If post-menopausal, subjects must have experienced at least 1 year of amenorrhea and provide a medical note from her physician documenting this medical history
* Agree not to travel to a malaria endemic area during the course of the study
* Agree to refrain from blood donation from the time of CHMI and for 3 years following CHMI
* Must be willing to take anti-malarial treatment after CHMI
* Must agree to stay in a pre-determined hotel near the NMRC CTC from approximately 7 days after CHMI until antimalarial treatment is completed or through 18 days post CHMI
* For active-duty military personnel, documentation of their command's approval to participate

Exclusion Criteria:

* Pregnant (positive urine pregnancy test) or nursing at screening or plans to become pregnant or nurse at any period from the time of enrollment through 56 days after CHMI.
* Receipt of any investigational malaria vaccine
* Any history of malaria infection
* Travel to a malaria endemic region within 6 months of enrollment or during the study (from enrollment through 2 months after CHMI)
* History of long-term residence (>5 years) in an area known to have significant transmission of P falciparum (http://www.cdc.gov/malaria/map/)
* History of clinically significant contact dermatitis
* Seropositive for the human immunodeficiency virus (HIV), hepatitis C virus (HCV), and/or hepatitis B surface antigen (HBsAg)
* Positive sickle cell screening test, including evidence of sickle cell trait or sickle cell anemia (due to its effect on subject's susceptibility to malaria)
* History of thalassemia or thalassemia trait (due to its effect on subject's susceptibility to malaria)
* Participation in any clinical study involving another investigational vaccine, drug, or other products within 60 days prior to enrollment or plan to participate in such a clinical study during or within 1 month following the active study phase of the study (from the day enrollment through 2 months after CHMI)
* Allergy to any component of the PfSPZ Challenge formulation, Malarone® (atovaquone-proguanil), and/or Coartem® (artemether-lumefantrine)
* History of porphyria

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 0 (Actual)
Dates: Start 2020-03 (Estimated); Primary Completion 2021-06 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Difference in the pre-patent period | 29 days
  The difference in the time of first malaria event (symptom or sign of malaria),in subjects infected with PfSPZ Challenge (NF54) vs. PfSPZ Challenge (7G8)
Difference in the total number of malaria events | 29 days
  The difference in the total number of Grade 2 or greater malaria events (symptoms and signs of malaria) experienced by subjects infected with PfSPZ Challenge (NF54) vs PfSPZ Challenge (7G8)

SECONDARY OUTCOMES:
Determine differences in pre-patent periods | 29 days
  Determine differences in prepatent periods in subjects infected with PfSPZ Challenge (NF54) vs PfSPZ Challenge (7G8) as detected by TBS, RDT, hsRDT and by PCR
Determine differences in the growth rate of parasites | 29 days
  Determine differences in the growth rate of parasites in the blood of subjects infected by PfSPZ Challenge (NF54) vs PfSPZ Challenge (7G8) as detected by PCR